CLINICAL TRIAL: NCT05978791
Title: Study on the Thrombolytic Effect of Platelet Membrane Coated Recombinant Staphylokinase on Human Arterial Thrombus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Director of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Other Study IDs: 021
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Arterial Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalized patients with suspected coronary artery disease: Take aspirin and ticagrelor maintenance dose ≥3 days, or loading dose of aspirin (300mg) and ticagrelor (180mg) ≥12 hours
  Interventions: Procedure: collection of venous blood or arterial blood
- healthy volunteers: Age 18-75 years old, body weight ≥45kg, regardless of gender;
  Interventions: Procedure: collection of venous blood or arterial blood

INTERVENTIONS:
Procedure: collection of venous blood or arterial blood — 1. Partial CAD patients were collected 20 mL arterial blood samples 12 hours after the last intake of 100mg aspirin and 2 hours after intake of 90mg ticagrelor. The blood samples were divided into 2 mL centrifuge tubes, with each containing 1.0 mL (for preparation of blood clots).
  2. Partial CAD patients were collected 40 mL blood samples into sodium citrate anticoagulant tubes 12 hours after the last intake of 100mg aspirin and 2 hours after intake of 90mg ticagrelor (for preparation of platelet-poor plasma, PPP).
  3. Healthy volunteer (group 1) collected 40 mL blood samples into sodium citrate anticoagulant tubes (for preparation of PPP).
  4. Healthy volunteer (group 2) collected 9 mL venous blood samples (for platelet aggregation assay).

SUMMARY:
Recombinant staphylokinase (r-SAK) is a third-generation thrombolytic agent produced by genetic engineering technology in 1985, which has better thrombolytic effect than streptokinase (SK) and urokinase (UK). It has similar biological properties to natural SAK, is highly selective to fibrin, does not activate systemic fibrinolysis, and can dissolve clots in a short period of time without significantly increasing the risk of bleeding, especially for platelet-rich arterial clots. Previous studies have shown that the thrombolytic revascularization rate of r-SAK is significantly better than that of r-SK and UK at the same dose in the rabbit model of acute femoral artery occlusive thrombosis. The revascularization rate of coronary artery at 90 minutes after thrombolysis was significantly higher with r-SAK than r-tPA. The combination of thrombolytic drugs and nanocarriers may provide a new solution for the existing thrombolytic therapy. Inspired by the natural affinity of platelets (PLT) in hemostasis and pathological thrombosis, we have developed a thrombus targeting nanocarrier, which is a platelet membrane cloaked r-SAK（PLT-SAK）and compare the thrombolytic effect of PLT-SAK with different doses of free r-SAK on human arterial thrombus, aiming to further improve the thrombolytic effectiveness of r-SAK.

DETAILED DESCRIPTION:
Currently, the most important treatment for thrombus and related cardiovascular diseases is prevention, but in the case of long-term thrombosis, the main treatment options include balloon catheters, surgical removal of embolus, thrombolytic therapy, and other related operations. Considering the cost of surgical treatment and its damage to the body, thrombolytic therapy has become one of the most effective ways to achieve rapid thrombus clearance and recanalization of blocked blood vessels in thrombotic diseases.

Recombinant staphylokinase (r-SAK) is a third-generation thrombolytic agent produced by genetic engineering technology in 1985, which has better thrombolytic effect than streptokinase (SK) and urokinase (UK). It has similar biological properties to natural SAK, is highly selective to fibrin, does not activate systemic fibrinolysis, and can dissolve clots in a short period of time without significantly increasing the risk of bleeding, especially for platelet-rich arterial clots. Previous studies have shown that the thrombolytic revascularization rate of r-SAK is significantly better than that of r-SK and UK at the same dose in the rabbit model of acute femoral artery occlusive thrombosis. The revascularization rate of coronary artery at 90 minutes after thrombolysis was significantly higher with r-SAK than r-tPA. The combination of thrombolytic drugs and nanocarriers may provide a new solution for the existing thrombolytic therapy. Inspired by the natural affinity of platelets (PLT) in hemostasis and pathological thrombosis, we have developed a thrombus targeting nanocarrier, which is a platelet membrane cloaked r-SAK（PLT-SAK）and compare the thrombolytic effect of PLT-SAK with different doses of free r-SAK on human arterial thrombus, aiming to further improve the thrombolytic effectiveness of r-SAK.

ELIGIBILITY:
For CAD patients:

Inclusion Criteria:

1. Age 18-75 years old, body weight ≥45kg, regardless of gender;
2. Patients with suspected coronary artery disease scheduled for coronary angiography or interventional therapy.
3. Take aspirin and ticagrelor maintenance dose ≥3 days, or loading dose of aspirin (300mg) and ticagrelor (180mg) ≥12 hours;

Exclusion Criteria:

1. Previous thrombolytic therapy with r-SAK;
2. A previous diagnosis of Staphylococcus aureus infection;
3. Those who are enrolled in other clinical trials;
4. Those who were deemed ineligible by other investigators.

For healthy volunteer:

Inclusion Criteria:

1. Age 18-75 years old, body weight ≥45kg, regardless of gender;

Exclusion Criteria:

1. Currently taking any medication that may affect platelet function, such as antiplatelet drugs or nonsteroidal anti-inflammatory drugs.
2. Individuals with blood disorders, active bleeding or a tendency to bleed, including platelet count <100×10^9/L, hemoglobin <100g/L, or recent bleeding in the digestive system or urinary tract within one month.
3. Individuals with impaired liver or kidney function, including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels above the upper limit of normal reference range, and estimated glomerular filtration rate (eGFR) <90 mL/min/1.73m^2 (calculated based on the CKD-EPI equation).
4. Recent (within one month) severe trauma, surgery, or head injury.
5. Pregnant or lactating women.
6. Diabetes.
7. Smokers.
8. Those who are enrolled in other clinical trials;
9. Those who were deemed ineligible by other investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. patients with suspected coronary artery disease scheduled for coronary angiography or interventional therapy；
  2. healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Thrombolysis rate | 60 min
  Thrombolysis rate (%) = [(initial clot weight - final clot weight) / initial clot weight] × 100%.

SECONDARY OUTCOMES:
Adenosine diphosphate-induced platelet aggregation rate. | 120 min
  9 mL venous blood was collected from healthy volunteers (group 2) into 3.2% sodium citrate tubes and subjected to platelet aggregation assay by light transmission aggregometry within 120min.Also test the effect of 20% aspirin- and ticagrelor-treated PPP and 20% healthy volunteers (group 1) PPP on platelet aggregation.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Background] Tillett WS, Garner RL. THE FIBRINOLYTIC ACTIVITY OF HEMOLYTIC STREPTOCOCCI. J Exp Med. 1933 Sep 30;58(4):485-502. doi: 10.1084/jem.58.4.485. PMID 19870210
- [Background] MACFARLANE RG, PILLING J. Fibrinolytic activity of normal urine. Nature. 1947 Jun 7;159(4049):779. doi: 10.1038/159779a0. No abstract available. PMID 20241608
- [Background] Rijken DC, Collen D. Purification and characterization of the plasminogen activator secreted by human melanoma cells in culture. J Biol Chem. 1981 Jul 10;256(13):7035-41. PMID 6787058
- [Background] Noble S, McTavish D. Reteplase. A review of its pharmacological properties and clinical efficacy in the management of acute myocardial infarction. Drugs. 1996 Oct;52(4):589-605. doi: 10.2165/00003495-199652040-00012. PMID 8891469
- [Background] Simpson D, Siddiqui MA, Scott LJ, Hilleman DE. Reteplase: a review of its use in the management of thrombotic occlusive disorders. Am J Cardiovasc Drugs. 2006;6(4):265-85. doi: 10.2165/00129784-200606040-00007. PMID 16913828
- [Background] Nordt TK, Bode C. Thrombolysis: newer thrombolytic agents and their role in clinical medicine. Heart. 2003 Nov;89(11):1358-62. doi: 10.1136/heart.89.11.1358. No abstract available. PMID 14594904
- [Background] Ross AM, Gao R, Coyne KS, Chen J, Yao K, Yang Y, Qin X, Qiao S, Yao M; TUCC Investigators. A randomized trial confirming the efficacy of reduced dose recombinant tissue plasminogen activator in a Chinese myocardial infarction population and demonstrating superiority to usual dose urokinase: the TUCC trial. Am Heart J. 2001 Aug;142(2):244-7. doi: 10.1067/mhj.2001.116963. PMID 11479462
- [Background] Gao RL, Han YL, Yang XC, Mao JM, Fang WY, Wang L, Shen WF, Li ZQ, Jia GL, Lu SZ, Wei M, Zeng DY, Chen JL, Qin XW, Xu B, DU CH; Collaborative Research Group of Reperfusion Therapy in Acute Myocardial Infarction (RESTART). Thorombolytic therapy with rescue percutaneous coronary intervention versus primary percutaneous coronary intervention in patients with acute myocardial infarction: a multicenter randomized clinical trial. Chin Med J (Engl). 2010 Jun;123(11):1365-72. PMID 20819587
- [Background] Nedaeinia R, Faraji H, Javanmard SH, Ferns GA, Ghayour-Mobarhan M, Goli M, Mashkani B, Nedaeinia M, Haghighi MHH, Ranjbar M. Bacterial staphylokinase as a promising third-generation drug in the treatment for vascular occlusion. Mol Biol Rep. 2020 Jan;47(1):819-841. doi: 10.1007/s11033-019-05167-x. Epub 2019 Nov 1. PMID 31677034
- [Background] Toombs CF. New directions in thrombolytic therapy. Curr Opin Pharmacol. 2001 Apr;1(2):164-8. doi: 10.1016/s1471-4892(01)00030-3. PMID 11714091
- [Background] Szemraj J, Stankiewicz A, Rozmyslowicz-Szerminska W, Mogielnicki A, Gromotowicz A, Buczko W, Oszajca K, Bartkowiak J, Chabielska E. A new recombinant thrombolytic and antithrombotic agent with higher fibrin affinity - a staphylokinase variant. An in-vivo study. Thromb Haemost. 2007 Jun;97(6):1037-45. doi: 10.1160/th06-10-0562. PMID 17549308
- [Background] Li CJ, Huang J, Yang ZJ, Cao KJ. Thrombolytic efficacy of native recombinant staphylokinase on femoral artery thrombus of rabbits. Acta Pharmacol Sin. 2007 Jan;28(1):58-65. doi: 10.1111/j.1745-7254.2007.00455.x. PMID 17184583
- [Background] Vanderschueren S, Barrios L, Kerdsinchai P, Van den Heuvel P, Hermans L, Vrolix M, De Man F, Benit E, Muyldermans L, Collen D, et al. A randomized trial of recombinant staphylokinase versus alteplase for coronary artery patency in acute myocardial infarction. The STAR Trial Group. Circulation. 1995 Oct 15;92(8):2044-9. doi: 10.1161/01.cir.92.8.2044. PMID 7554180
- [Background] Kamaly N, Yameen B, Wu J, Farokhzad OC. Degradable Controlled-Release Polymers and Polymeric Nanoparticles: Mechanisms of Controlling Drug Release. Chem Rev. 2016 Feb 24;116(4):2602-63. doi: 10.1021/acs.chemrev.5b00346. Epub 2016 Feb 8. PMID 26854975
- [Background] Shen S, Wu Y, Liu Y, Wu D. High drug-loading nanomedicines: progress, current status, and prospects. Int J Nanomedicine. 2017 May 31;12:4085-4109. doi: 10.2147/IJN.S132780. eCollection 2017. PMID 28615938
- [Background] Tan YF, Lao LL, Xiong GM, Venkatraman S. Controlled-release nanotherapeutics: State of translation. J Control Release. 2018 Aug 28;284:39-48. doi: 10.1016/j.jconrel.2018.06.014. Epub 2018 Jun 15. PMID 29902484
- [Background] Tietjen GT, Bracaglia LG, Saltzman WM, Pober JS. Focus on Fundamentals: Achieving Effective Nanoparticle Targeting. Trends Mol Med. 2018 Jul;24(7):598-606. doi: 10.1016/j.molmed.2018.05.003. Epub 2018 Jun 5. PMID 29884540
- [Background] Falati S, Gross P, Merrill-Skoloff G, Furie BC, Furie B. Real-time in vivo imaging of platelets, tissue factor and fibrin during arterial thrombus formation in the mouse. Nat Med. 2002 Oct;8(10):1175-81. doi: 10.1038/nm782. Epub 2002 Sep 16. PMID 12244306
- [Background] Lippi G, Franchini M, Targher G. Arterial thrombus formation in cardiovascular disease. Nat Rev Cardiol. 2011 Jul 5;8(9):502-12. doi: 10.1038/nrcardio.2011.91. PMID 21727917
- [Background] Hu CM, Fang RH, Wang KC, Luk BT, Thamphiwatana S, Dehaini D, Nguyen P, Angsantikul P, Wen CH, Kroll AV, Carpenter C, Ramesh M, Qu V, Patel SH, Zhu J, Shi W, Hofman FM, Chen TC, Gao W, Zhang K, Chien S, Zhang L. Nanoparticle biointerfacing by platelet membrane cloaking. Nature. 2015 Oct 1;526(7571):118-21. doi: 10.1038/nature15373. Epub 2015 Sep 16. PMID 26374997
- [Background] Cheng JW, Zhang XJ, Cheng LS, Li GY, Zhang LJ, Ji KX, Zhao Q, Bai Y. Low-Dose Tissue Plasminogen Activator in Acute Ischemic Stroke: A Systematic Review and Meta-Analysis. J Stroke Cerebrovasc Dis. 2018 Feb;27(2):381-390. doi: 10.1016/j.jstrokecerebrovasdis.2017.09.014. Epub 2017 Oct 27. PMID 29111341
- [Background] Zamanlu M, Farhoudi M, Eskandani M, Mahmoudi J, Barar J, Rafi M, Omidi Y. Recent advances in targeted delivery of tissue plasminogen activator for enhanced thrombolysis in ischaemic stroke. J Drug Target. 2018 Feb;26(2):95-109. doi: 10.1080/1061186X.2017.1365874. Epub 2017 Aug 25. PMID 28796540
- [Background] Ma YH, Liu CH, Liang Y, Chen JP, Wu T. Targeted Delivery of Plasminogen Activators for Thrombolytic Therapy: An Integrative Evaluation. Molecules. 2019 Sep 19;24(18):3407. doi: 10.3390/molecules24183407. PMID 31546842
- [Background] Hassanpour S, Kim HJ, Saadati A, Tebon P, Xue C, van den Dolder FW, Thakor J, Baradaran B, Mosafer J, Baghbanzadeh A, de Barros NR, Hashemzaei M, Lee KJ, Lee J, Zhang S, Sun W, Cho HJ, Ahadian S, Ashammakhi N, Dokmeci MR, Mokhtarzadeh A, Khademhosseini A. Thrombolytic Agents: Nanocarriers in Controlled Release. Small. 2020 Oct;16(40):e2001647. doi: 10.1002/smll.202001647. Epub 2020 Aug 12. PMID 32790000